CLINICAL TRIAL: NCT00699387
Title: Population Pharmacokinetics Study of Benznidazole in Children With Chagas Disease
Brief Title: Population Pharmacokinetics of Benznidazole in Children With Chagas Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Collaborators: Thrasher Research Fund (Other); The Hospital for Sick Children (Other); Fundacion Bunge y Born (Argentina) (Unknown); Universidad Nacional de La Plata (Other); Consejo de Investigacion en Salud Gobierno de Buenos Aires (Other)
Responsible Party: Dr Jaime Altcheh, Servicio de Parasitología, Hospital de Niños "R Gutiérrez" de Buenos Aires
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHAGAS-CHILDREN-POPPK
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Chagas Disease
Keywords: Chagas disease; Pediatrics; benznidazole; population pharmacokinetics; neglected diseases; parasitology; pediatric clinical pharmacology
MeSH Terms: conditions — Chagas Disease; Neglected Diseases | interventions — benzonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Benznidazole (Experimental): Treatment of pediatric Chagas disease with benznidazole
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: Benznidazole — benznidazole (RADANIL®, Roche) 5-8 mg/kg/d bid PO for 60 days
  Other Names: Children with Chagas Disease Treated with Benznidazole; Niños con Chagas en Tratamiento con Benznidazol

SUMMARY:
Background: Chagas disease is a parasitic infection caused by the Trypanosome cruzi. The initial phase of the infection happens mainly in children. Up to 10% of infected children die. Survivors often develop chronic infection leading to heart disease and other complications in 30% of patients. These complications often result in death or severe handicaps in early adulthood, depriving societies of individuals in their most productive years.

There are 20 million people infected in Latin America. Complications lead to 20,000 deaths every year.

Treatment during the acute phase with benznidazole leads to a high cure rate. However, there are very few studies of this drug and virtually none in children, even though benznidazole was developed over 30 years ago.

Hypotheses and Specific Aims: We hypothesize that the pharmacokinetics of benznidazole in children is different from adults, and that obtaining information on how it is absorbed, distributed and eliminated in children will allow optimization of treatment of Chagas disease in this population. This will in turn improve the outlook for children by reducing mortality and long term complications. We aim to study the pharmacokinetics of benznidazole in children receiving the drug for treatment of Chagas disease, and to correlate it with treatment effectiveness and incidence of adverse effects.

Potential Impact: This novel knowledge will allow better and more rational approaches to the treatment of Chagas disease. It will also set the foundation for further studies that will be able to test improved therapies that may increase treatment response in vulnerable children.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 - 12 years old of both sexes, with a diagnosis of Chagas' disease and eligible for treatment with benznidazole, as per current treatment protocols.
* Chagas disease diagnostic criteria: At least 2 positive serological tests for Trypanosoma cruzi infection (ELISA, hemoagglutination, particle agglutination tests).
* Informed consent signed by the parents, and consent or assent of the patients (according to age and consenting capacity).

Exclusion Criteria:

* Patients with a history of hypersensitivity to benznidazole or any of the drug excipients
* Immunocompromised patients
* Altered hepatic function (increase in AST/ALT x3 or bilirubin x3) or altered renal function (increase in creatinine x3)
* Pregnancy

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Description of Population pharmacokinetics parameters of benznidazole (i.e. median population clearance, absorption and volume of distribution, and their respective inter-individual variabilities) | 2 months (treatment period)

SECONDARY OUTCOMES:
Adverse events | 2 months (treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Altcheh, MD, Study Director — Parasitology Service, Children's Hospital "R. Gutierrez" of Buenos Aires; Facundo Garcia Bournissen, MD, Principal Investigator — Division of Clinical Pharmacology & Toxicology, Hospital for Sick Children, University of Toronto; Norberto Giglio, MD, Principal Investigator — Epidemiology Service, Children's Hospital "R. Gutierrez" of Buenos Aires; Gideon Koren, MD, Principal Investigator — Division of Clinical Pharmacology &Toxicology, Hospital for Sick Children, University of Toronto; Oscar Della Vedova, Principal Investigator — Universidad Nacional de La Plata; Guido Mastrantonio, Principal Investigator — Facultad de Ciencias Exactas, Universidad Nacional de La Plata
Locations (1):
- Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Altcheh J, Moscatelli G, Mastrantonio G, Moroni S, Giglio N, Marson ME, Ballering G, Bisio M, Koren G, Garcia-Bournissen F. Population pharmacokinetic study of benznidazole in pediatric Chagas disease suggests efficacy despite lower plasma concentrations than in adults. PLoS Negl Trop Dis. 2014 May 22;8(5):e2907. doi: 10.1371/journal.pntd.0002907. eCollection 2014 May. PMID 24853169